CLINICAL TRIAL: NCT03809663
Title: A Dose-Ranging, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Tezepelumab Alone or Combined With Topical Corticosteroids in Moderate-to-Severe Atopic Dermatitis
Brief Title: A Dose Ranging Placebo-Controlled Double-Blind Study to Evaluate the Safety and Efficacy of Tezepelumab in Atopic Dermatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Tezepelumab as a monotherapy in atopic dermatitis did not reach the targeted efficacy level pre-established for this patient population.
Sponsor: Amgen (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20170755; 2018-001997-52 (EudraCT Number)
Record Dates: First submitted 2019-01-10; First posted 2019-01-18 (Actual); Results first posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; eczema; tezepelumab; dermatology; dermatitis; inflammation; skin; moderate dermatitis; severe dermatitis
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Dermatitis; Inflammation | interventions — tezepelumab

STUDY DESIGN:
Intervention Model Description: This phase 2b study is designed to evaluate the safety and efficacy of tezepelumab as a monotherapy and explore its efficacy as adjunct therapy in subjects with moderate-to-severe AD. This study consists of Part A (the main study evaluating tezepelumab as a monotherapy) and Part B (a study evaluating tezepelumab as adjunctive therapy when combined with a topical corticosteroid regimen
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A: Placebo (Placebo Comparator): Matching placebo administered via SC injection Q2W for a maximum of 52 weeks.
  Participants defined as non-responders (those who do not achieve at least 50% improvement in EASI at Week 16 compared to baseline) will switch to receive tezepelumab 420 mg SC injection Q2W for the remainder of the study beginning with the Week 18 dose.
  Interventions: Other: Placebo
- Part A: Tezepelumab 210 mg (Experimental): Tezepelumab 210 mg administered via SC injection once every 4 weeks (Q4W) from Week 4 for a maximum of 52 weeks.
  All participants randomized to tezepelumab will receive 420 mg SC injection as their first dose. Participants will then receive a placebo at Week 2 to maintain blinding.
  Participants defined as non-responders (those who do not achieve at least 50% improvement in EASI at Week 16 compared to baseline) will switch to receive tezepelumab 420 mg SC injection Q2W for the remainder of the study beginning with the Week 18 dose.
  Interventions: Drug: Tezepelumab
- Part A: Tezepelumab 280 mg (Experimental): Tezepelumab 280 mg administered via SC injection Q2W from Week 2 for a maximum of 52 weeks.
  All participants randomized to tezepelumab will receive 420 mg SC injection as their first dose. Participants will then receive their randomized dose of 280 mg Q2W from Week 2.
  Participants defined as non-responders (those who did not achieve at least 50% improvement in EASI at Week 16 compared to baseline) will switch to receive tezepelumab 420 mg SC injection Q2W for the remainder of the study beginning with the Week 18 dose.
  Interventions: Drug: Tezepelumab
- Part A: Tezepelumab 420 mg (Experimental): Tezepelumab 420 mg administered via SC injection Q2W for a maximum of 52 weeks.
  Interventions: Drug: Tezepelumab
- Part B: Placebo and Topical Corticosteroids Regimen (Experimental): Matching placebo administered via SC injection Q2W with topical corticosteroids (TCS) for a maximum of 52 weeks.
  Interventions: Drug: Tezepelumab
- Part B: Tezepelumab 420 mg and Topical Corticosteroids Regimen (Experimental): Tezepelumab 420 mg administered via SC injection Q2W with TCS for a maximum of 52 weeks.
  Interventions: Drug: Tezepelumab

INTERVENTIONS:
Drug: Tezepelumab — Solution for injection
  Other Names: AMG157
  Arms: Part A: Tezepelumab 210 mg; Part A: Tezepelumab 280 mg; Part A: Tezepelumab 420 mg; Part B: Placebo and Topical Corticosteroids Regimen; Part B: Tezepelumab 420 mg and Topical Corticosteroids Regimen
Other: Placebo — Placebo solution for injection
  Arms: Part A: Placebo

SUMMARY:
This phase 2b study is designed to evaluate the safety and efficacy of tezepelumab as a monotherapy and explore its efficacy as adjunct therapy in subjects with moderate-to-severe atopic dermatitis (AD).

DETAILED DESCRIPTION:
All subjects will receive a subcutaneous (SC) dose of either investigational product or placebo as the first dose on day 1.

Subjects who are determined to be non-responders in Part A will receive tezepelumab SC every 2 weeks (Q2W) following completion of all week 16 study activities. Nonresponders are defined as those subjects who have not achieved at least a 50% improvement in Eczema Area and Severity Index (EASI) at week 16 compared to baseline (day 1).

Safety follow-up is 18 weeks after the end of treatment (EOT) visit (20 weeks after the final dose of investigational product).

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent prior to initiation of any study specific activities/procedures.
* Age greater than or equal to 18 to less than or equal to 75 years at screening.
* Clinical diagnosis of chronic AD (also known as atopic eczema) for at least 2 years prior to screening and has confirmed AD (Hanifin and Rajka criteria for AD (Hanifin and Rajka, 1980).
* AD that affects greater than or equal to' 10% body surface area as assessed by EASI at screening and on day 1.
* An IGA score of greater than or equal to 3 at screening and on day 1.
* An EASI score of greater than or equal to 16 at screening and on day 1.
* Subject discontinued treatment with TCS, topical calcineurin inhibitors (TCI), and prescription moisturizers containing TCS or topical calcineurin inhibitors (TCI) for at least the 7 days immediately prior to the first dose of investigational product
* Documented recent history (within 12 months before the screening visit) of inadequate response totreatment with topical TCS or subjects for whom topical treatments are otherwise medically inadvisable (ie, because of important side effects or safety risks).

  * Inadequate response is defined as failure to achieve and maintain remission or a low disease activity state (comparable to IGA 0 = clear to IGA 2 = mild) despite treatment with a daily regimen of TCS of medium or higher potency (with or without TCI as appropriate).

Exclusion Criteria:

* Active dermatologic conditions, which might confound the diagnosis of AD or would interfere with the assessment of treatment, such as scabies, seborrheic dermatitis, cutaneous lymphoma, ichthyosis, psoriasis, allergic contact dermatitis, or irritant contact dermatitis.
* History of a clinically significant infection within 28 days prior to day 1 that, in the opinion of the investigator or medical monitor, might compromise the safety of the subject in the study, interfere with evaluation of the investigational product, or reduce the subject's ability to participate in the study. Clinically significant infections are defined as either of the following: 1) a systemic infection; or 2) a serious skin infection requiring parenteral antibiotic, antiviral, or antifungal medication.
* Diagnosis of a helminth parasitic infection within 6 months prior to screening that had not been treated with or had failed to respond to standard of care therapy.
* Documented medical history of chronic alcohol or drug abuse within 12 months prior to screening.
* History of anaphylaxis following any biologic therapy.
* Evidence of active liver disease at screening, including jaundice or aspartate aminotransferase (AST), alanine aminotransferase (ALT), or alkaline phosphatase greater than twice the upper limit of normal (ULN).
* Subjects who, in the opinion of the investigator, have evidence of active tuberculosis (TB), either treated or untreated, or a positive QuantiFERON-tuberculosis Gold (QFT-G) test for TB during screening. Subjects with an indeterminate QFT-G may be enrolled if they have ALL of the following:

  * No symptoms of TB: productive, prolonged cough (> 3 weeks); coughing up blood; fever; night sweats; unexplained appetite loss; unintentional weight loss
  * No evidence of active TB on chest radiograph within 3 months prior to the first dose of investigational product. Note: Chest radiograph is not part of screening procedure and will be the responsibility
* Positive hepatitis B surface antigen or hepatitis C antibody serology. Subjects with a history of hepatitis B vaccination without a history of hepatitis B are allowed to enroll in the study.
* Positive human immunodeficiency virus (HIV) test at screening or the subject is taking antiretroviral medications, as determined by medical history, prior medications, and/or the subject's verbal report.
* Other Medical Conditions>
* History of malignancy, except for basal cell carcinoma or in situ carcinoma of the cervix treated with apparent success with curative therapy ≥ 12 months prior to screening or other malignancies treated with apparent success with curative therapy ≥ 5 years prior to screening.
* History or evidence of severe depression, schizophrenia, previous suicide attempts, or suicidal ideation.

Prior/Concomitant Therapy:

* Subjects who are unwilling to abstain from the use of TCS, TCI, and prescription moisturizers (those that contain TCS and TCI) from screening through week 16 (applies only to Part A subjects)
* Subjects who have had side effects of topical medications including intolerance to treatment, hypersensitivity reactions, significant skin atrophy, or systemic effects as assessed by the investigator or by the subject's treating physician (applies only to Part B subjects)
* More than or equal to 30% of the total lesional surface is located on areas of thin skin that cannot be safely treated with medium or higher potency TCS (eg, face, neck, intertriginous areas, areas of skin atrophy) (applies only to Part B subjects)
* Receipt of any approved biologic agent (eg, dupilumab) within 4 months or 5 elimination half-lives (whichever is longer) prior to screening
* Have used immunosuppressive/immunomodulating drugs (eg, systemic corticosteroids, cyclosporine, mycophenolate-mofetil, interferon (IFN)-gamma, Janus kinase inhibitors, azathioprine, methotrexate) within 4 weeks prior to screening, or any condition that, in the opinion of the investigator, is likely to require such treatment(s) during the first 4 weeks of study treatment.
* Have had phototherapy for AD in the 2 months prior to day 1, and subjects unwilling to avoid phototherapy during the first 16 weeks of the study
* If on allergen-specific immunotherapy, subjects must be on a maintenance dose and schedule for ≥ 28 days prior to screening. Allergen-specific immunotherapy is defined as SC immunotherapy to aeroallergens and/o venom (Hymenoptera) as well as sublingual immunotherapy to aeroallergens
* Vaccination with a live or attenuated vaccine within 28 days prior to day 1. Receipt of inactive/killed vaccinations (eg, inactive influenza) is allowed. Note that receipt of the Th2 cytokine inhibitor suplatast within 15 days prior to randomization and during the study is not allowed.
* Major surgery within 8 weeks prior to screening or planned inpatient surgery or hospitalization during the study period
* Currently receiving treatment in another investigational device or drug study, or less than 6 months since ending treatment on another investigational device or drug study(ies). Other investigational procedures while participating in this study are excluded.

Other Exclusions:

* Female subject is pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 16 weeks after the last dose of investigational product. (Females of childbearing potential should only be enrolled in the study after a negative highly sensitive serum pregnancy test).
* Female subjects of childbearing potential who are sexually active with unsterilized male partners unwilling to use 1 highly effective method of contraception during treatment and for an additional 16 weeks after the last dose of investigational product. Cessation of contraception after this point must be discussed with a responsible physician. Females of childbearing potential are defined as those who are not surgically sterile (ie, had bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal (defined as 12 months with no menses without an alternative medical cause). A highly effective method of contraception is defined as one that resulted in a low failure rate (ie, < 1% per year) when used consistently and correctly.
* Subject has known sensitivity to any of the products or components to be administered during dosing.
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2020-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (86):
- United States (16):
  - First OC Dermatology, Fountain Valley, California
  - Clinical Science Institute, Santa Monica, California
  - Hamilton Research, LLC, Alpharetta, Georgia
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Dundee Dermatology, West Dundee, Illinois
  - DS Research, Clarksville, Indiana
  - Epiphany Dermatology of Kansas, LLC, Overland Park, Kansas
  - Skin Sciences Pllc, Louisville, Kentucky
  - Scott Health Services LLC, Louisville, Kentucky
  - Clarkston Skin Research, Clarkston, Michigan
  - J Woodson Dermatology and Associates, Henderson, Nevada
  - Mount Sinai Hospital, New York, New York
  - DermResearch Center of New York Inc, Stony Brook, New York
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Modern Research Associates, Dallas, Texas
  - Premier Clinical Research, Spokane, Washington
- Australia (5):
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - Veracity Clinical Research, Woolloongabba, Queensland
  - Skin Health Institute, Carlton, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Fremantle Dermatology, Fremantle, Western Australia
- Canada (7):
  - Doctor Chih-Ho Hong Medical Incorporated, Surrey, British Columbia
  - DermEffects, London, Ontario
  - Lynderm Research Inc, Markham, Ontario
  - Cheema Research Incorporated, Mississauga, Ontario
  - SKDS Research Incorporated, Newmarket, Ontario
  - Gordon Sussman Clinical Research Incorporated, North York, Ontario
  - JRB Research Incorporated, Ottawa, Ontario
- Czechia (5):
  - Fakultni nemocnice u sv Anny v Brne, Brno
  - Nemocnice Novy Jicin as, Nový Jičín
  - Fakultni nemocnice Ostrava, Ostrava-Poruba
  - Sanatorium profesora Arenbergera, Prague
  - Nemocnice Na Bulovce, Prague
- Estonia (3):
  - North Estonia Medical Centre, Tallinn
  - Clinical Research Centre, Tartu
  - Tartu University Hospital, Tartu
- Germany (3):
  - CharitÃ© Berlin, Berlin
  - UniversitÃ¤tsmedizin GÃ¶ttingen - Georg-August-UniversitÃ¤t, GÃ¶ttingen
  - Medizinische Hochschule Hannover, Hanover
- Hungary (6):
  - Csalogany Orvosi Kozpont, Budapest
  - Obudai Egeszsegugyi Centrum Kft, Budapest
  - Debreceni Egyetem Kenezy Gyula Egyetemi Korhaz, Debrecen
  - CRU Hungary Kft, Miskolc
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont Altalanos Orvostudomanyi Kar, Szeged
- Japan (12):
  - Toho University Sakura Medical Center, Sakura-shi, Chiba
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Takagi Dermatological Clinic, Obihiro-shi, Hokkaido
  - Medical Corporation Kojinkai Sapporo Skin Clinic, Sapporo, Hokkaido
  - Meiwa Hospital, Nishinomiya-shi, Hyōgo
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Kume Clinic, Sakai-shi, Osaka
  - Nippon Medical School Hospital, Bunkyo-ku, Tokyo
  - Japan Post Holdings Co Ltd Tokyo Teishin Hospital, Chiyoda-ku, Tokyo
  - NTT Medical Center Tokyo, Shinagawa-ku, Tokyo
  - Center Hospital of the National Center for Global Health and Medicine, Shinjuku-ku, Tokyo
  - Shirasaki Dermatology Clinic, Takaoka-shi, Toyama
- Latvia (4):
  - Riga First Hospital, Riga
  - J Kisis, Riga
  - Clinic Latvian Dermatology Institute, Riga
  - Outpatient Clinic of Ventspils, Ventspils
- Poland (8):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Centrum Terapii Wspolczesnej J M Jasnorzewska Spolka Komandytowo-Akcyjna, Lodz
  - Dermoklinika Centrum Medyczne Spolka cywilna M Kierstan J Narbutt A Lesiak, Lodz
  - Niepubliczny Zaklad Opieki Zdrowotnej Med Laser Borzecki Spolka Jawna, Lublin
  - Tomasz Blicharski Lubelskie Centrum Diagnostyczne, Świdnik
  - Centrum Medyczne Pratia Warszawa, Warsaw
  - Medicus Sp z o o, Wroclaw
  - DermMedica Spzoo, Wroclaw
- Hallym University Kangnam Sacred Heart Hospital, Seoul, South Korea
- Spain (6):
  - Hospital Universitario Virgen Macarena, Seville, AndalucÃ-a
  - Hospital Universitari Germans Trias i Pujol, Badalona, CataluÃ±a
  - Hospital del Mar, Barcelona, CataluÃ±a
  - Hospital de la Santa Creu i Sant Pau, Barcelona, CataluÃ±a
  - Hospital General Universitario de Alicante, Alicante, Valencia
  - Hospital Universitario de La Princesa, Madrid
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- Ukraine (6):
  - Chernivtsi Regional Skin and Venereal Dispensary, Chernivtsi
  - Regional Skin and Venereal Dispensary, Dnipro
  - Ivano-Frankivsk Regional Skin and Venereal Dispensary, Ivano-Frankivsk
  - Medical clinic Blagomed, Kyiv
  - Asclepius, Uzhhorod
  - Military Hospital, Military Unit A3309 of the Military Medical Clinical Center, Zaporizhzhia
- United Kingdom (3):
  - Ninewells Hospital, Dundee
  - Whipps Cross University Hospital, London
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in 78 centers in 14 countries including Australia, Canada, Czech Republic, Estonia, Germany, Hungary, Japan, Latvia, Poland, Republic of Korea, Spain, Ukraine, the United Kingdom, and the United States.
Pre-assignment Details: Enrollment of Part A of this study was completed as of 27 July 2020. The study was terminated prior to the enrollment of any participants into Part B.
Groups:
- Part A: Placebo: Matching placebo administered via subcutaneous (SC) injection once every 2 weeks (Q2W) for a maximum of 52 weeks.
  Participants defined as non-responders (those who did not achieve at least 50% improvement in Eczema Area and Severity Index [EASI] compared to baseline) at Week 16 switched to receive tezepelumab 420 mg SC injection Q2W for the remainder of the study.
- Part A: Tezepelumab 210 mg Q4W: Tezepelumab 210 mg administered via SC injection once every 4 weeks (Q4W) from Week 4 for a maximum of 52 weeks.
  All participants randomized to tezepelumab received 420 mg SC injection as their first dose. Participants then received a placebo at Week 2 and every other week to maintain blinding.
  Participants defined as non-responders (those who did not achieve at least 50% improvement in EASI compared to baseline) at Week 16 switched to receive tezepelumab 420 mg SC injection Q2W for the remainder of the study.
- Part A: Tezepelumab 280 mg Q2W: Tezepelumab 280 mg administered via SC injection Q2W from Week 2 for a maximum of 52 weeks.
  All participants randomized to tezepelumab received 420 mg SC injection as their first dose. Participants then received their randomized dose of 280 mg Q2W from Week 2.
  Participants defined as non-responders (those who did not achieve at least 50% improvement in EASI compared to baseline) at Week 16 switched to receive tezepelumab 420 mg SC injection Q2W for the remainder of the study.
- Part A: Tezepelumab 420 mg Q2W: Tezepelumab 420 mg administered via SC injection Q2W for a maximum of 52 weeks.
  Participants defined as non-responders (those who did not achieve at least 50% improvement in EASI compared to baseline) at Week 16 stayed to receive tezepelumab 420 mg SC injection Q2W for the remainder of the study.
- Part B: Placebo and Topical Corticosteroids Regimen: Matching placebo was planned to be administered via SC injection Q2W with topical corticosteroids (TCS) for a maximum of 52 weeks.
  The study was terminated prior to the start of Part 2 and no participants were enrolled.
- Part B: Tezepelumab 420 mg Q2W and Topical Corticosteroids Regimen: Tezepelumab 420 mg was planned to be administered via SC injection Q2W with TCS for a maximum of 52 weeks.
  The study was terminated prior to the start of Part 2 and no participants were enrolled.
Period: Overall Study
Arm/Group | Part A: Placebo | Part A: Tezepelumab 210 mg Q4W | Part A: Tezepelumab 280 mg Q2W | Part A: Tezepelumab 420 mg Q2W | Part B: Placebo and Topical Corticosteroids Regimen | Part B: Tezepelumab 420 mg Q2W and Topical Corticosteroids Regimen
Started | 63 | 62 | 63 | 63 | 0 | 0
Participants Who Received Investigational Product | 63 | 61 | 63 | 63 | 0 | 0
EASI 50 Non-responder at Week 16 | 40 | 26 | 30 | 38 | 0 | 0
Switched to Tezepelumab 420 mg Q2W After Week 16 | 39 | 24 | 30 | 38 | 0 | 0
Completed | 12 | 18 | 15 | 16 | 0 | 0
Not Completed | 51 | 44 | 48 | 47 | 0 | 0
Not completed — Decision by sponsor | 24 | 18 | 20 | 20 | 0 | 0
Not completed — Withdrawal by Subject | 26 | 22 | 27 | 26 | 0 | 0
Not completed — Lost to Follow-up | 1 | 4 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): All randomized participants in Part A.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Placebo | Part A: Tezepelumab 210 mg Q4W | Part A: Tezepelumab 280 mg Q2W | Part A: Tezepelumab 420 mg Q2W | Total
Number analyzed (Participants) | 63 | 62 | 63 | 63 | 251
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.7 (13.4) | 38.5 (15.0) | 36.9 (13.4) | 40.7 (14.3) | 37.9 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 32 | 23 | 27 | 109
  Male | 36 | 30 | 40 | 36 | 142
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 1 | 4 | 15
  Not Hispanic or Latino | 57 | 58 | 62 | 59 | 236
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 21 | 16 | 16 | 13 | 66
  Black or African-American | 1 | 3 | 1 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  White | 41 | 42 | 45 | 47 | 175
  Unknown | 0 | 0 | 0 | 0 | 0
  Other | 0 | 0 | 1 | 0 | 1
Investigator's Global Assessment Score [Count of Participants; unit: Participants] — The IGA allows investigators to assess overall disease severity at 1 given time point and consists of a 6-point severity scale from clear to severe disease
  * 0 = clear
  * 1 = almost clear
  * 2 = mild disease
  * 3 = moderate disease
  * 4 = severe disease
  * 5 = very severe disease The IGA uses clinical characteristics of erythema, infiltration, papulation, oozing & crusting as guidelines for the overall severity assessment (Breuer et al 2004).
  Participants
    IGA Score of 3 | 26 | 37 | 26 | 37 | 126
    IGA Score of 4 | 32 | 17 | 30 | 18 | 97
    IGA Score of 5 | 5 | 8 | 7 | 8 | 28
Eczema Area and Severity Index (EASI) [Mean (Standard Deviation); unit: Score on a scale] — The EASI was designed by modifying the Psoriasis Area and Severity Index (Schmitt et al, 2007). The EASI evaluates 4 natural anatomical regions for severity and extent of key disease signs and focuses on key acute and chronic signs of inflammation (ie, erythema, induration/papulation, excoriation, and lichenification).
  The lowest possible total score is 0 and the highest possible total score is 72, with higher scores indicating greater severity of eczema.
  Score on a scale | 32.0 (11.1) | 28.4 (13.2) | 30.3 (10.7) | 28.6 (12.4) | 29.8 (11.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Investigator's Global Assessment (IGA) Score of 0 (Clear) or 1 (Almost Clear) (IGA 0/1) at Week 16
Description: The IGA allows investigators to assess overall disease severity at 1 given time point and consists of a 6-point severity scale from clear to severe disease
  * 0 = clear
  * 1 = almost clear
  * 2 = mild disease
  * 3 = moderate disease
  * 4 = severe disease
  * 5 = very severe disease
  The IGA uses clinical characteristics of erythema, infiltration, papulation, oozing, and crusting as guidelines for the overall severity assessment (Breuer et al, 2004).
  Participants who took rescue medication between Day 29 to Week 16 were considered non-responders.
Time Frame: Week 16
Population: FAS: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: Tezepelumab 210 mg Q4W | Part A: Tezepelumab 280 mg Q2W | Part A: Tezepelumab 420 mg Q2W
Number analyzed (Participants) | 63 | 62 | 63 | 63
Participants | 2 | 4 | 2 | 5
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Tezepelumab 210 mg Q4W; Test type: Superiority; p = 0.56, Regression, Logistic — Nominal p-value; Odds Ratio (OR) = 1.686, 95% CI 2-sided [0.290 to 9.809]
Statistical Analysis 2: Comparison: Part A: Placebo vs Part A: Tezepelumab 280 mg Q2W; Test type: Superiority; p = 0.99, Regression, Logistic — Nominal p-value; Odds Ratio (OR) = 1.011, 95% CI 2-sided [0.135 to 7.551]
Statistical Analysis 3: Comparison: Part A: Placebo vs Part A: Tezepelumab 420 mg Q2W; Test type: Superiority; p = 0.38, Regression, Logistic — Nominal p-value; Odds Ratio (OR) = 2.146, 95% CI 2-sided [0.390 to 11.800]

2. Primary Outcome: Number of Participants Who Experienced a 75% Reduction From Baseline in Eczema Area and Severity Index (EASI 75) at Week 16
Description: The EASI evaluates 4 natural anatomical regions for severity and extent of key disease signs and focuses on key acute and chronic signs of inflammation (ie, erythema, induration/papulation, excoriation, and lichenification).
  A reduction in the EASI score indicates an improvement in severity. Participants who took rescue medication between Day 29 to Week 16 were considered non-responders.
Time Frame: Baseline and Week 16
Population: FAS: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: Tezepelumab 210 mg Q4W | Part A: Tezepelumab 280 mg Q2W | Part A: Tezepelumab 420 mg Q2W
Number analyzed (Participants) | 63 | 62 | 63 | 63
Participants | 8 | 9 | 10 | 7
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Tezepelumab 210 mg Q4W; Test type: Superiority; p = 0.97, Regression, Logistic — Nominal p-value; Odds Ratio (OR) = 0.982, 95% CI 2-sided [0.344 to 2.803]
Statistical Analysis 2: Comparison: Part A: Placebo vs Part A: Tezepelumab 280 mg Q2W; Test type: Superiority; p = 0.70, Regression, Logistic — Nominal p-value; Odds Ratio (OR) = 1.217, 95% CI 2-sided [0.441 to 3.356]
Statistical Analysis 3: Comparison: Part A: Placebo vs Part A: Tezepelumab 420 mg Q2W; Test type: Superiority; p = 0.58, Regression, Logistic — Nominal p-value; Odds Ratio (OR) = 0.730, 95% CI 2-sided [0.243 to 2.197]

3. Secondary Outcome: Number of Participants Who Experienced a 50% or 90% Reduction From Baseline in Eczema Area and Severity Index (EASI 50/90) at Week 16
Description: as for outcome 2
Time Frame: Baseline and Week 16
Population: FAS: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: Tezepelumab 210 mg Q4W | Part A: Tezepelumab 280 mg Q2W | Part A: Tezepelumab 420 mg Q2W
Number analyzed (Participants) | 56 | 58 | 58 | 56
Participants
  EASI 50 | 11 | 21 | 18 | 11
  EASI 90 | 3 | 3 | 3 | 3

4. Secondary Outcome: Time to Achievement of 50%, 75% or 90% Reduction From Day 1 in Eczema Area and Severity Index (EASI 50/75/90)
Time Frame: Day 1 up to End of Study Visit (Week 70)
Population: FAS: All randomized participants.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Part A: Placebo | Part A: Tezepelumab 210 mg Q4W | Part A: Tezepelumab 280 mg Q2W | Part A: Tezepelumab 420 mg Q2W
Number analyzed (Participants) | 63 | 62 | 63 | 63
Weeks
  Time to EASI 50 | 6.143 [4.14 to 19.57] | 8.143 [3.86 to 16.14] | 6.286 [3.86 to 22.14] | 5.857 [3.86 to 16.14]
  Time to EASI 75 | 6.143 [4.14 to 19.57] | 6.286 [4.00 to 16.43] | 6.714 [4.14 to 22.14] | 6.429 [4.14 to 16.14]
  Time to EASI 90 | 8.286 [4.43 to 19.57] | 10.929 [4.00 to 16.14] | 10.071 [6.14 to 16.14] | 7.286 [4.14 to 16.29]

5. Secondary Outcome: Change From Baseline in Scoring of Atopic Dermatitis (SCORAD) at Week 16
Description: The SCORAD is a clinical tool for assessing the severity (ie, extent, intensity) of atopic dermatitis (AD). The tool evaluates the extent and intensity of the AD lesions, along with subjective symptoms (Kunz et al, 1997). The total score ranges from 0 to 103, with higher values indicating more severe disease. A negative change from baseline indicates an improvement in severity of disease.
Time Frame: Baseline and Week 16
Population: FAS: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Part A: Placebo | Part A: Tezepelumab 210 mg Q4W | Part A: Tezepelumab 280 mg Q2W | Part A: Tezepelumab 420 mg Q2W
Number analyzed (Participants) | 63 | 62 | 63 | 63
Score on a scale | -8.00 (2.55) | -16.75 (2.40) | -11.87 (2.49) | -9.32 (2.48)

6. Secondary Outcome: Change From Baseline in Pruritus Numeric Rating Scale (NRS) at Week 16
Description: Pruritus was assessed using an NRS (0-10) with 0 = no itch and 10 = worst imaginable itch. A negative change from baseline indicates an improvement in symptoms.
Time Frame: Baseline and Week 16
Population: FAS: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Part A: Placebo | Part A: Tezepelumab 210 mg Q4W | Part A: Tezepelumab 280 mg Q2W | Part A: Tezepelumab 420 mg Q2W
Number analyzed (Participants) | 63 | 62 | 63 | 63
Score on a scale | -0.71 (0.30) | -1.40 (0.27) | -0.94 (0.28) | -0.38 (0.28)

7. Secondary Outcome: Serum Trough Concentrations of Tezepelumab After Q2W or Q4W Administration
Description: Switchers were included up to Week 16 and were then excluded from the analysis after switching. All Tezepelumab participants received 420 mg of Tezepelumab on Day 1.
Time Frame: Pre-dose on Day 1, Week 2, 4, 12, 16, 24, 32, 40, 48, 50, 52, 58 and 70
Population: All randomized participants who received at least 1 dose of investigational product with analyzable samples at each time point. Participants were analyzed according to the highest dose of actual treatment received after initial first dose or only dose received. Switchers were included up to Week 16 and were then excluded from the analysis after switching at Week 16.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Part A: Tezepelumab 210 mg Q4W | Part A: Tezepelumab 280 mg Q2W | Part A: Tezepelumab 420 mg Q2W
Number analyzed (Participants) | 58 | 58 | 66
µg/mL
  Day 1 | 0.00031 (0.00236) | 0.00 (0.00) | 0.00 (0.00)
  Week 2: number analyzed (Participants) | 51 | 49 | 60
  Week 2 | 34.9 (10.9) | 36.3 (12.9) | 34.8 (12.9)
  Week 4: number analyzed (Participants) | 56 | 48 | 53
  Week 4 | 23.4 (9.03) | 48.8 (16.0) | 58.9 (21.4)
  Week 12: number analyzed (Participants) | 49 | 48 | 47
  Week 12 | 21.7 (8.47) | 66.7 (22.9) | 97.0 (35.0)
  Week 16: number analyzed (Participants) | 47 | 46 | 44
  Week 16 | 22.2 (9.42) | 77.4 (33.0) | 98.0 (37.8)
  Week 24: number analyzed (Participants) | 20 | 17 | 11
  Week 24 | 23.2 (10.6) | 83.6 (31.2) | 107 (29.5)
  Week 32: number analyzed (Participants) | 16 | 15 | 5
  Week 32 | 25.4 (17.0) | 75.1 (36.3) | 81.4 (26.4)
  Week 40: number analyzed (Participants) | 11 | 6 | 4
  Week 40 | 22.9 (12.7) | 76.8 (19.7) | 112 (63.3)
  Week 48: number analyzed (Participants) | 5 | 5 | 5
  Week 48 | 18.2 (6.49) | 76.4 (26.4) | 118 (48.3)
  Week 50: number analyzed (Participants) | 5 | 4 | 4
  Week 50 | 29.2 (9.11) | 86.8 (27.7) | 113 (44.4)
  Week 52: number analyzed (Participants) | 4 | 5 | 4
  Week 52 | 18.3 (7.24) | 67.2 (33.2) | 102 (31.2)
  Week 58: number analyzed (Participants) | 3 | 3 | 2
  Week 58 | 5.41 (2.56) | 18.0 (7.09) | 20.9 (NA) — Insufficient samples to measure standard deviation.
  Week 70: number analyzed (Participants) | 4 | 3 | 3
  Week 70 | 0.699 (0.380) | 1.87 (1.74) | 5.36 (3.20)

8. Secondary Outcome: Serum Trough Concentrations of Tezepelumab After Switching to 420 mg Q2W Administration After Week 16
Time Frame: Pre-dose on Week 24, 32, 40, 48, 50, 52, 58 and 70
Population: All randomized participants who received at least 1 dose of investigational product who were assessed as EASI non-responders at Week 16 and switched to 420 mg Q2W, with analyzable samples at each time point.
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- Part A: Placebo up to Week 16; Tezepelumab 420 mg Week 16 to 52 (Switchers): All participants who received the matching placebo Q2W up to Week 16 and were assessed as EASI 50 non-responders and switched to receive tezepelumab 420 mg Q2W up to Week 52.
  Tezepelumab 420 mg administered via SC injection Q2W from Week 18 to Week 52.
- Part A: Tezepelumab 210 mg up to Week 16; Tezepelumab 420 mg Week 16 to 52 (Switchers): All participants who received tezepelumab 210 mg Q4W up to Week 16 and were assessed as EASI 50 non-responders and switched to receive tezepelumab 420 mg Q2W up to Week 52 (switchers).
  Tezepelumab 420 mg administered via SC injection Q2W from Week 18 to Week 52.
- Part A: Tezepelumab 280 mg up to Week 16; Tezepelumab 420 mg Week 16 to 52 (Switchers): All participants who received tezepelumab 280 mg Q2W up to Week 16 and were assessed as EASI 50 non-responders and switched to receive tezepelumab 420 mg Q2W up to Week 52 (switchers).
  Tezepelumab 420 mg administered via SC injection Q2W from Week 18 to Week 52.
- Part A: Tezepelumab 420 mg up to Week 16; Tezepelumab 420 mg Week 16 to 52 (Switchers): All participants who received tezepelumab 420 mg Q2W up to Week 16 and were assessed as EASI 50 non-responders and continued to receive tezepelumab 420 mg Q2W up to Week 52.
  Tezepelumab 420 mg administered via SC injection Q2W from Week 18 to Week 52.
Arm/Group | Part A: Placebo up to Week 16; Tezepelumab 420 mg Week 16 to 52 (Switchers) | Part A: Tezepelumab 210 mg up to Week 16; Tezepelumab 420 mg Week 16 to 52 (Switchers) | Part A: Tezepelumab 280 mg up to Week 16; Tezepelumab 420 mg Week 16 to 52 (Switchers) | Part A: Tezepelumab 420 mg up to Week 16; Tezepelumab 420 mg Week 16 to 52 (Switchers)
Number analyzed (Participants) | 30 | 22 | 21 | 25
µg/mL
  Week 24 | 70.5 (28.3) | 87.2 (24.0) | 96.6 (29.2) | 100 (38.2)
  Week 32: number analyzed (Participants) | 23 | 15 | 17 | 24
  Week 32 | 91.0 (38.7) | 104 (38.8) | 97.8 (39.3) | 105 (39.1)
  Week 40: number analyzed (Participants) | 15 | 11 | 9 | 15
  Week 40 | 117 (42.7) | 93.8 (35.5) | 113 (31.1) | 101 (37.7)
  Week 48: number analyzed (Participants) | 9 | 6 | 5 | 9
  Week 48 | 134 (60.2) | 121 (29.1) | 89.6 (35.1) | 103 (29.9)
  Week 50: number analyzed (Participants) | 10 | 5 | 5 | 8
  Week 50 | 115 (39.0) | 125 (42.2) | 79.1 (38.6) | 106 (27.0)
  Week 52: number analyzed (Participants) | 9 | 6 | 4 | 8
  Week 52 | 125 (30.8) | 113 (45.0) | 88.3 (33.0) | 105 (30.2)
  Week 58: number analyzed (Participants) | 4 | 1 | 1 | 4
  Week 58 | 26.0 (21.6) | 52.6 (NA) — Insufficient number of samples to calculate standard deviation. | 36.7 (NA) — Insufficient number of samples to calculate standard deviation. | 17.6 (9.28)
  Week 70: number analyzed (Participants) | 9 | 5 | 4 | 7
  Week 70 | 5.07 (5.10) | 4.47 (3.39) | 2.60 (1.72) | 3.49 (2.42)

ADVERSE EVENTS:
Time Frame: Up to week 16 for Arms 1-4 and after week 16 up to week 70 for Arms 5-12
Description: Other Adverse Events include all non-serious events that occurred at a frequency of greater than or equal to 5 percent.
Groups:
- Placebo: Participants who took placebo from Week 1 to Week 16.
- Tezepelumab 210 mg Q4W: Participants who took 210 mg Q4W from Week 1 to Week 16.
- Tezepelumab 280 mg Q2W: Participants who took 280 mg Q2W from Week 1 to Week 16.
- Tezepelumab 420 mg Q2W: Participants who took 420 mg Q2W from Week 1 to Week 16.
  Includes 7 subjects randomized to the lower doses of Tezepelumab but received only the first dose of Tezepelumab 420 mg SC and early discontinued.
- Placebo - Placebo: Non-switching participants who took placebo from Week 16 to Week 52.
- Tezepelumab 210 mg Q4W - 210 mg Q4W: Non-switching participants who took 210 mg Q4W from Week 16 to Week 52.
- Tezepelumab 280 mg Q2W - 280 mg Q2W: Non-switching participants who took 280 mg Q2W from Week 16 to Week 52.
- Tezepelumab 420 mg Q2W - 420 mg Q2W: Non-switching participants who continued to take 420 mg Q2W from Week 16 to Week 52.
  Includes 6 participants who were randomized to placebo (n=2), 210 mg Q4W (n=3) and 280 mg Q2W (n=1) but switched to Tezepelumab 420 mg SC Q2W in error after Week 16.
- Placebo- Tezepelumab 420 mg Q2W; Tezepelumab 210 mg Q4W-420 mg Q2W; Tezepelumab 280 mg Q2W-420 mg Q2W: Participants who switched after Week 16 to take 420 mg Q2W.
- Tezepelumab 420 mg Q2W-420 mg Q2W: Participants who switched after week 16 who continued to take 420 mg Q2W.
Arm/Group | Placebo | Tezepelumab 210 mg Q4W | Tezepelumab 280 mg Q2W | Tezepelumab 420 mg Q2W | Placebo - Placebo | Tezepelumab 210 mg Q4W - 210 mg Q4W | Tezepelumab 280 mg Q2W - 280 mg Q2W | Tezepelumab 420 mg Q2W - 420 mg Q2W | Placebo- Tezepelumab 420 mg Q2W | Tezepelumab 210 mg Q4W-420 mg Q2W | Tezepelumab 280 mg Q2W-420 mg Q2W | Tezepelumab 420 mg Q2W-420 mg Q2W
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/59 | 0/58 | 0/70 | 0/12 | 0/25 | 0/20 | 0/22 | 0/39 | 0/24 | 0/30 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/63 | 2/59 | 0/58 | 1/70 | 0/12 | 0/25 | 1/20 | 0/22 | 2/39 | 0/24 | 1/30 | 4/38
Other Adverse Events (participants affected / at risk) | 25/63 | 20/59 | 29/58 | 30/70 | 6/12 | 10/25 | 11/20 | 5/22 | 18/39 | 9/24 | 10/30 | 19/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=63) | Tezepelumab 210 mg Q4W (N=59) | Tezepelumab 280 mg Q2W (N=58) | Tezepelumab 420 mg Q2W (N=70) | Placebo - Placebo (N=12) | Tezepelumab 210 mg Q4W - 210 mg Q4W (N=25) | Tezepelumab 280 mg Q2W - 280 mg Q2W (N=20) | Tezepelumab 420 mg Q2W - 420 mg Q2W (N=22) | Placebo- Tezepelumab 420 mg Q2W (N=39) | Tezepelumab 210 mg Q4W-420 mg Q2W (N=24) | Tezepelumab 280 mg Q2W-420 mg Q2W (N=30) | Tezepelumab 420 mg Q2W-420 mg Q2W (N=38)
Corneal degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Device failure (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dermatitis herpetiformis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=63) | Tezepelumab 210 mg Q4W (N=59) | Tezepelumab 280 mg Q2W (N=58) | Tezepelumab 420 mg Q2W (N=70) | Placebo - Placebo (N=12) | Tezepelumab 210 mg Q4W - 210 mg Q4W (N=25) | Tezepelumab 280 mg Q2W - 280 mg Q2W (N=20) | Tezepelumab 420 mg Q2W - 420 mg Q2W (N=22) | Placebo- Tezepelumab 420 mg Q2W (N=39) | Tezepelumab 210 mg Q4W-420 mg Q2W (N=24) | Tezepelumab 280 mg Q2W-420 mg Q2W (N=30) | Tezepelumab 420 mg Q2W-420 mg Q2W (N=38)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chalazion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Application site pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Condition aggravated (General disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Temperature intolerance (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Food allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Eczema herpeticum (Infections and infestations) | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Herpes zoster (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 6 | 5 | 10 | 6 | 0 | 3 | 3 | 3 | 3 | 0 | 3 | 3
Oral herpes (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pharyngitis (Infections and infestations) | 3 | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Pyoderma (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 3 | 2 | 1 | 0 | 1 | 2 | 0 | 2 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
SARS-CoV-2 antibody test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 3 | 1 | 1 | 4 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 12 | 9 | 13 | 13 | 2 | 5 | 2 | 3 | 9 | 2 | 4 | 6
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin striae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 3 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Enrollment of Part A of this study was completed as of 27 July 2020. The study was terminated prior to the enrollment of any participants into Part B.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/63/NCT03809663/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT03809663/SAP_001.pdf